CLINICAL TRIAL: NCT03529058
Title: Evaluation of Hypophosphatemia as a Predictive Marker of Mortality During Sepsis in ICU
Brief Title: Hypophosphatemia as a Predictive Marker of Mortality During Sepsis in ICU
Acronym: PORPOISE-REA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PORPOISE-REA ( 29BRC17.0180)
Record Dates: First submitted 2018-04-05; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2017-11

CONDITIONS: Hypophosphatemia; Infection
MeSH Terms: conditions — Hypophosphatemia; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study in the 3 intensive care units of the Brest Teaching Hospital (France) during a 18-months period (June 2014 -December 2015) to study the independent association between hypophosphatemia and 90-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Blood stream infection

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to 21-bed medical ICU, 15-bed surgical ICU and 8-bed cardiothoracic ICU between June 1, 2014 and December 31, 2015 were screened for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
90-day mortality | 90 days since the first blood stream infection in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

REFERENCES:
- [Derived] Padelli M, Aubron C, Huet O, Hery-Arnaud G, Vermeersch V, Hoffmann C, Bettacchioli E, Maguet H, Carre JL, Leven C. Is hypophosphataemia an independent predictor of mortality in critically ill patients with bloodstream infection? A multicenter retrospective cohort study. Aust Crit Care. 2021 Jan;34(1):47-54. doi: 10.1016/j.aucc.2020.05.001. Epub 2020 Jul 27. PMID 32732023